CLINICAL TRIAL: NCT03067428
Title: Effects of Fructose Restriction on Liver Steatosis
Acronym: FRUITLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 162034
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Nonalcoholic Fatty Liver Disease; Glucose Metabolism Disorders; Endothelial Dysfunction
Keywords: Fructose; Diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Glucose Metabolism Disorders | interventions — Glucose; Fructose

STUDY DESIGN:
Intervention Model Description: double blind, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose (Active Comparator): Participants will follow a six-week low fructose diet. The amount of restricted fructose will be supplemented as glucose powder.
  Interventions: Dietary Supplement: Glucose
- Fructose (Placebo Comparator): Participants will follow a six-week low fructose diet. The amount of restricted fructose will be supplemented as fructose powder.
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Glucose — Participants will adhere to a fructose restricted diet for a period of six weeks (<7.5 grams/meal and/or <10 grams/day; ad-libitum intake). In addition, the amount of fructose that will be restricted - which is based on the average individual fructose intake assessed prior to randomization - will be supplemented as glucose powder three times daily during the meal.
  Arms: Glucose
Dietary Supplement: Fructose — Participants will adhere to a fructose restricted diet for a period of six weeks (<7.5 grams/meal and/or <10 grams/day; ad-libitum intake). In addition, the amount of fructose that will be restricted - which is based on the average individual fructose intake assessed prior to randomization - will be supplemented as fructose powder three times daily during the meal.
  Arms: Fructose

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is an emerging health problem as it can lead to end stage liver failure and cardiovascular complications. Diet play an important role in the development of NAFLD. Many studies have addressed the effects of added fructose on NAFLD. To date, little attention has been paid to the effects of a diet devoid of fructose. Therefore, the investigators aim to study the effects of fructose restriction on hepatic fat accumulation and vascular function using a double-blind randomized placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index ≥ 28 kg/m2
* Fatty liver index ≥ 60
* Fructose intake ≥45 grams/day

Exclusion Criteria:

* Medical history of liver disease
* (History of) excessive alcohol consumption (defined as > 2 units/day for women, and > 3 units/day for men)
* Major change in weight and/or physical activity prior to the study
* Use of glucose lowering drugs
* Recent illness
* Pregnancy and/or lactation
* Contraindications for magnetic resonance imaging
* Inability to give informed consent

Protocol change (implemented on July 18, 2018): in order to increase the inclusion of study participants, subjects with an average daily fructose intake < 45 gram/day will also be eligible for participation. In subjects who have an average daily fructose intake < 45 gram/day, supplementation of either fructose or glucose (see 'Arms and Interventions') will be increased to 45 gram/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in intrahepatic triglyceride content | 6 weeks
  Assessed by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Change in arterial stiffness (PWV) | 6 weeks
  Assessed by pulse wave velocity
Change in endothelial function (flowmotion and skin heating response) | 6 weeks
  Assessed by laser doppler flowmetry
Change in endothelial function (RHI) | 6 weeks
  Assessed by reactive hyperemia peripheral arterial tonometry
Change in endothelial function (panel of endothelial dysfunction biomarkers) | 6 weeks
  Assessed by plasma biomarkers
Change in glucose metabolism | 6 weeks
  Assessed by a standard 75-gram oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Martijn CG Brouwers, MD,PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Simons PIHG, Simons N, van de Waarenburg MPH, Bons JAP, van der Ploeg EMC, Feskens EJM, Schalkwijk CG, Brouwers MCGJ. Effects of glucose and fructose supplementation on serum sex hormone-binding globulin and testosterone levels: Post-hoc analysis of a double-blind randomized controlled trial. Clin Nutr ESPEN. 2025 Oct;69:384-388. doi: 10.1016/j.clnesp.2025.07.1123. Epub 2025 Jul 26. PMID 40721209
- [Derived] Janssen LEF, Simons N, Simons PIHG, Schaper NC, Feskens EJM, van der Ploeg LMC, Van den Eynde MDG, Schalkwijk CG, Houben AJHM, Stehouwer CDA, Brouwers MCGJ. Effects of fructose restriction on blood pressure: Secondary analysis of a double-blind randomized controlled trial. Clin Nutr ESPEN. 2022 Oct;51:97-103. doi: 10.1016/j.clnesp.2022.07.009. Epub 2022 Jul 30. PMID 36184254
- [Derived] Simons N, Veeraiah P, Simons PIHG, Schaper NC, Kooi ME, Schrauwen-Hinderling VB, Feskens EJM, van der Ploeg EMCL, Van den Eynde MDG, Schalkwijk CG, Stehouwer CDA, Brouwers MCGJ. Effects of fructose restriction on liver steatosis (FRUITLESS); a double-blind randomized controlled trial. Am J Clin Nutr. 2021 Feb 2;113(2):391-400. doi: 10.1093/ajcn/nqaa332. PMID 33381794